CLINICAL TRIAL: NCT00053482
Title: The Effect of Dose on Safety, Tolerability, and Immunogenicity of ACAM2000 Smallpox Vaccine in Adults With Previous Smallpox Vaccination
Brief Title: Dose Study of ACAM2000 Smallpox Vaccine in Previously Vaccinated Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emergent BioSolutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-400-003
Record Dates: First submitted 2003-01-30; First posted 2003-01-31 (Estimated); Results first posted 2011-02-11 (Estimated); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Smallpox
Keywords: Smallpox vaccines; Dryvax®; Orthopoxvirus; Vaccinia virus; ACAM2000
MeSH Terms: conditions — Smallpox; Vaccinia | interventions — ACAM2000; DryVax vaccine; Smallpox Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group 1: ACAM2000 (Experimental): Participants will receive dose 1 of the ACAM2000 smallpox vaccine
  Interventions: Biological: ACAM2000 Smallpox Vaccine
- Group 2: ACAM2000 (Experimental): Participants will receive dose 2 of the ACAM2000 smallpox vaccine
  Interventions: Biological: ACAM2000 Smallpox Vaccine
- Group 3: ACAM2000 (Experimental): Participants will receive dose 3 of the ACAM2000 smallpox vaccine
  Interventions: Biological: ACAM2000 Smallpox Vaccine
- Group 4: ACAM2000 (Experimental): Participants will receive dose 4 of the ACAM2000 smallpox vaccine
  Interventions: Biological: ACAM2000 Smallpox Vaccine
- Group 5: Dryvax® (Active Comparator): Participants will receive dose 1 of Dryvax® smallpox vaccine.
  Interventions: Biological: Vaccinia virus (calf lymph) smallpox vaccine: Dryvax®

INTERVENTIONS:
Biological: ACAM2000 Smallpox Vaccine — Group 1 dose: 1.0x10-8th PFU/ml, Group 2 dose: 2.0x10-7th PFU/ml, Group 3 dose: 1.0x10-7th PFU/ml, Group 4 dose: 5.0x10-6th PFUL/ml
  Arms: Group 1: ACAM2000; Group 2: ACAM2000; Group 3: ACAM2000; Group 4: ACAM2000
Biological: Vaccinia virus (calf lymph) smallpox vaccine: Dryvax® — Group 5 dose: 1.0x10-8th PFU/ml
  Other Names: Dryvax®
  Arms: Group 5: Dryvax®

SUMMARY:
The objective of this study is to determine the minimum dose of ACAM2000 needed to produce a cutaneous reaction in at least 90% of a population of healthy adults at least 28 years of age and previously vaccinated against smallpox.

DETAILED DESCRIPTION:
Specifically, the objectives of this study are to:

1. Compare the safety and tolerability of four dose levels of ACAM2000 and a standard dose of Dryvax® in healthy adults at least 28 years of age and previously vaccinated to smallpox. Safety and tolerability will be determined by examination of the local cutaneous reaction, adverse events, physical examinations, vital signs, structured interviews, and laboratory analysis.
2. Determine the immunogenicity of four dose levels of ACAM2000 and a standard dose of Dryvax® in healthy adults at least 28 years of age by comparing:

   1. the proportion of subjects at each dose level who develop a major cutaneous reaction
   2. the proportion of subjects in each treatment group who develop neutralizing antibodies, including the fold-increase in antibody titer between Baseline and Day 30 sera; and the geometric mean vaccinia neutralizing antibody titer on Day 30.
3. Determine the minimum dose of ACAM2000 that is calculated to produce a major cutaneous reaction in at least 90% of a population of healthy adults at least 28 years of age, with a history of smallpox vaccination.

ELIGIBILITY:
Inclusion criteria:

* have a history of previous smallpox vaccination greater than 10 years previous to the date of screening and presence of a vaccination scar.
* females must not be pregnant, lactating and must agree to use an effective form of birth control for the 30 days following vaccination or unable to bear children.
* agree to be available for the entire study and agree to comply with all requirements.

exclusion criteria:

* children 1 year of age or younger in the household or be in close contact
* smallpox vaccination within ten years
* known or suspected Human immunodeficient virus (HIV) infection, primary immunodeficiency disorder, leukemia, lymphoma, or current radiation treatment or use of immunosuppressive or anti-neoplastic drugs or have a household member or intimate contact with the conditions listed above.
* renal disease
* current or past history of eczema or a household member or direct contact who has eczema.
* known allergy or past allergic reactions to latex gloves or to antibiotics which include neomycin, streptomycin, chlortetracycline, and polymyxin B
* known allergy or past allergic reaction to blood products.
* known allergy to cidofovir or sulfa-containing drugs.
* history of allergic phenomena following smallpox vaccination in the past, including urticaria, erythema multiforme, or Stevens-Johnson syndrome.
* transfusion of blood or treatment with any blood product.
* current or history of drug or alcohol abuse
* innoculation with any other live vaccine or participating in another drug or vaccine trial within 30 days of enrollment.

Min Age: 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2003-01; Primary Completion 2003-04 (Actual); Study Completion 2003-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Emergent BioSolutions
Locations (3):
- United States (3):
  - PRA International, Lenexa, Kansas
  - Bio-Kinetic Clinical Applications, Springfield, Missouri
  - Memorial Hospital of Rhode Island Division of Infectious Diseases, Pawtucket, Rhode Island

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 07 January 2003 to 31 March 2003 in 3 medical centers in the US.
Pre-assignment Details: A total of 357 participants who met the inclusion and exclusion criteria were enrolled and vaccinated.
Groups:
- ACAM2000 Dose 1: Participants received a single dose of ACAM2000 smallpox vaccine, 1.0x10-8th plaque-forming units/mL on Day 0
- ACAM2000 Dose 2: Participants received a single dose of ACAM2000 smallpox vaccine, 2.0x10-7th plaque-forming units/mL on Day 0
- ACAM2000 Dose 3: Participants received a single dose of ACAM2000 smallpox vaccine, 1.0x10-7th plaque-forming units/mL on Day 0
- ACAM2000 Dose 4: Participants received a single dose of ACAM2000 smallpox vaccine, 5.0x10-6th plaque-forming units/mL on Day 0
- Dryvax® Vaccine: Participants received a single dose of Dryvax® smallpox vaccine, 1.0x10-8th plaque-forming units/mL on Day 0
Period: Overall Study
Arm/Group | ACAM2000 Dose 1 | ACAM2000 Dose 2 | ACAM2000 Dose 3 | ACAM2000 Dose 4 | Dryvax® Vaccine
Started | 51 | 102 | 102 | 50 | 52
Completed | 51 | 102 | 102 | 50 | 52
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ACAM2000 Dose 1 | ACAM2000 Dose 2 | ACAM2000 Dose 3 | ACAM2000 Dose 4 | Dryvax® Vaccine | Total
Number analyzed (Participants) | 51 | 102 | 102 | 50 | 52 | 357
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 51 | 102 | 102 | 50 | 52 | 357
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48 (9.7) | 48 (10.1) | 50 (11.7) | 47 (9.1) | 48 (9.2) | 48 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 57 | 54 | 18 | 19 | 175
  Male | 24 | 45 | 48 | 32 | 33 | 182
Region of Enrollment [Number; unit: participants]
  United States | 51 | 102 | 102 | 50 | 52 | 357

OUTCOME MEASURES:

1. Primary Outcome: The Neutralizing Antibody Response Titers Post-vaccination With ACAM2000 or Dryvax® Smallpox Vaccine
Description: The neutralizing antibody response titers were determined by the Plaque-Reduction Neutralization Test (PRNT50)
Time Frame: Day 30 post-vaccination
Population: The neutralizing antibody response titers were assessed in the antibody evaluable, per-protocol population.
Measure: Mean (Standard Deviation); unit: PRNT50 Titers
Arm/Group | ACAM2000 Dose 1 | ACAM2000 Dose 2 | ACAM2000 Dose 3 | ACAM2000 Dose 4 | Dryvax® Vaccine
Number analyzed (Participants) | 51 | 102 | 102 | 50 | 52
PRNT50 Titers
  Baseline | 77 (119.4) | 112 (280.5) | 76 (108.7) | 91 (145.4) | 186 (709.8)
  Day 15 | 244 (485.4) | 259 (449.1) | 802 (4111.6) | 546 (829.9) | 1287 (2198.4)

2. Primary Outcome: Participants With ≥ 4-fold Increase in Plaque-Reduction Neutralization Test (PRNT50) Titers Post-vaccination With ACAM2000 or Dryvax® Smallpox Vaccine.
Time Frame: Day 30 post-vaccination
Measure: Number; unit: Participants
Arm/Group | ACAM2000 Dose 1 | ACAM2000 Dose 2 | ACAM2000 Dose 3 | ACAM2000 Dose 4 | Dryvax® Vaccine
Number analyzed (Participants) | 51 | 102 | 102 | 50 | 52
Participants | 13 | 31 | 41 | 38 | 39

3. Primary Outcome: Number of Participants Reporting Adverse Events of Severe Intensity Post-vaccination With ACAM2000 or Dryvax® Smallpox Vaccine
Time Frame: Days 0 to 30 post-vaccination
Population: Post-vaccination adverse events were assessed in the safety, intent-to-treat population.
Measure: Number; unit: Participants
Arm/Group | ACAM2000 Dose 1 | ACAM2000 Dose 2 | ACAM2000 Dose 3 | ACAM2000 Dose 4 | Dryvax® Vaccine
Number analyzed (Participants) | 51 | 102 | 102 | 50 | 52
Participants
  Lymph Node Pain | 1 | 1 | 1 | 1 | 0
  Lymphadenopathy | 0 | 0 | 1 | 0 | 0
  Constipation | 0 | 0 | 1 | 0 | 0
  Toothache | 0 | 1 | 0 | 0 | 0
  Injection Site Erythema | 0 | 1 | 3 | 4 | 3
  Injection Site Pruritus | 0 | 1 | 0 | 0 | 1
  Injection Site Pain | 0 | 0 | 0 | 0 | 1
  Human Immunodeficiency Virus (HIV) Test Positive | 1 | 0 | 0 | 0 | 0
  Back Pain | 0 | 1 | 0 | 0 | 0
  Myalgia | 1 | 0 | 0 | 0 | 0
  Swelling Not Otherwise Specified | 0 | 0 | 0 | 1 | 0
  Migraine Not Otherwise Specified | 0 | 1 | 0 | 0 | 0
  Pregnancy Not Otherwise Specified | 0 | 1 | 0 | 0 | 0
  Calculus Renal Not Otherwise Specified | 0 | 1 | 0 | 0 | 0

4. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Rash Events Post-vaccination With ACAM2000 or Dryvax® Smallpox Vaccine
Time Frame: Days 0 to 30 post-vaccination
Population: Treatment-emergent rash events were assessed in the safety intent-to-treat population.
Measure: Number; unit: Participants
Arm/Group | ACAM2000 Dose 1 | ACAM2000 Dose 2 | ACAM2000 Dose 3 | ACAM2000 Dose 4 | Dryvax® Vaccine
Number analyzed (Participants) | 51 | 102 | 102 | 50 | 52
Participants
  Rash Not Otherwise Specified | 2 | 5 | 5 | 5 | 3
  Rash Macular | 0 | 0 | 0 | 1 | 0
  Rash Papular | 0 | 0 | 1 | 0 | 0
  Application Site Rash | 0 | 0 | 1 | 1 | 2
  Injection Site Rash | 1 | 0 | 1 | 0 | 2
  Any Rash | 3 | 5 | 8 | 7 | 5

5. Other Pre Specified Outcome: Selected Hematology Parameters (Hematocrit, Lymphocyte, and Eosinophil) at Baseline and Day 15 Post-vaccination With ACAM2000 or Dryvax® Smallpox Vaccine
Time Frame: Days 0 (Baseline) and 15 post-vaccination
Population: The hematology parameters were assessed in the intent-to-treat safety population.
Measure: Mean (Standard Deviation); unit: Percentage (%)
Arm/Group | ACAM2000 Dose 1 | ACAM2000 Dose 2 | ACAM2000 Dose 3 | ACAM2000 Dose 4 | Dryvax® Vaccine
Number analyzed (Participants) | 51 | 102 | 102 | 50 | 52
Percentage (%)
  Hematocrit (Baseline) | 41.7 (3.58) | 42.4 (3.87) | 42.2 (3.66) | 42.8 (3.69) | 43.3 (3.62)
  Hematocrit (Day15) | 41.2 (3.53) | 41.6 (3.86) | 41.5 (3.68) | 42.1 (3.30) | 42.8 (3.27)
  Lymphocytes (Baseline) | 31.8 (7.27) | 30.8 (6.68) | 30.6 (7.87) | 30.4 (6.98) | 30.9 (6.27)
  Lymphocytes (Day15) | 32.4 (6.88) | 30.8 (7.19) | 31.3 (8.26) | 31.2 (7.36) | 33.4 (7.00)
  Eosinophils (Baseline) | 2.8 (1.89) | 2.5 (2.09) | 2.5 (1.50) | 2.3 (1.37) | 2.8 (1.84)
  Eosinophils (Day15) | 2.5 (1.43) | 2.5 (2.02) | 2.6 (1.66) | 2.5 (1.55) | 3.1 (2.2)

6. Other Pre Specified Outcome: Selected Hematology Parameters (Red Bood Cell and Platelets) at Baseline and Day 15 Post-vaccination With ACAM2000 or Dryvax® Smallpox Vaccine
Time Frame: Days 0 (Baseline) and 15 post-vaccination
Population: The hematology parameters were assessed in the intent-to-treat safety population.
Measure: Mean (Standard Deviation); unit: x10^6th/µL
Arm/Group | ACAM2000 Dose 1 | ACAM2000 Dose 2 | ACAM2000 Dose 3 | ACAM2000 Dose 4 | Dryvax® Vaccine
Number analyzed (Participants) | 51 | 102 | 102 | 50 | 52
x10^6th/µL
  Red Blood Cell count (Baseline) | 4.7 (0.35) | 4.8 (0.47) | 4.8 (0.46) | 4.9 (0.40) | 4.9 (0.45)
  Red Blood Cell count (Day15) | 4.7 (0.36) | 4.7 (0.50) | 4.7 (0.50) | 4.8 (0.36) | 4.8 (0.41)
  Platelets (Baseline) | 279 (69.7) | 276 (54.5) | 277 (71.5) | 285 (58.4) | 280 (75.7)
  Platelets (Day15) | 286 (66.7) | 281 (61.3) | 276 (67.2) | 284 (63.2) | 284 (77.0)

7. Other Pre Specified Outcome: Clinical Chemistry Parameters (Creatinine and Glucose) at Baseline and Day 15 Post-vaccination With ACAM2000 or Dryvax® Smallpox Vaccine
Time Frame: Days 0 (Baseline) and 15 post-vaccination
Population: Clinical chemistry parameters were assessed in the intent-to-treat safety population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | ACAM2000 Dose 1 | ACAM2000 Dose 2 | ACAM2000 Dose 3 | ACAM2000 Dose 4 | Dryvax® Vaccine
Number analyzed (Participants) | 51 | 102 | 102 | 50 | 52
mg/dL
  Creatinine (Baseline) | 0.90 (0.122) | 0.94 (0.167) | 0.92 (0.187) | 0.94 (0.184) | 0.97 (0.156)
  Creatinine (Day 15) | 0.91 (0.145) | 0.96 (0.181) | 0.95 (0.184) | 0.96 (0.184) | 0.98 (0.138)
  Glucose (Baseline) | 91 (11.7) | 87 (8.7) | 92 (15.3) | 92 (13.4) | 88 (10.7)
  Glucose (Day 15) | 94 (22.6) | 90 (18.9) | 90 (16.3) | 94 (28.4) | 95 (27.3)

8. Other Pre Specified Outcome: Clinical Chemistry Parameters (Aspartate Transaminase and Alanine Transaminase) at Baseline and Day 15 Post-vaccination With ACAM2000 or Dryvax® Smallpox Vaccine
Time Frame: Days 0 (Baseline) and 15 post-vaccination
Population: Clinical chemistry parameters were assessed in the intent-to-treat safety population
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | ACAM2000 Dose 1 | ACAM2000 Dose 2 | ACAM2000 Dose 3 | ACAM2000 Dose 4 | Dryvax® Vaccine
Number analyzed (Participants) | 51 | 102 | 102 | 50 | 52
IU/L
  Aspartate transaminase (Baseline) | 27 (13.2) | 24 (9.9) | 23 (10.3) | 22 (6.9) | 22 (6.2)
  Aspartate transaminase (Day 15) | 24 (11.5) | 23 (8.7) | 24 (10.7) | 21 (10.4) | 21 (5.8)
  Alanine transaminase (Baseline) | 39 (16.3) | 39 (19.5) | 37 (17.3) | 37 (15.7) | 36 (12.9)
  Alanine transaminase (Day 15) | 39 (20.1) | 38 (20.4) | 37 (19.2) | 37 (16.0) | 34 (13.8)

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the day of vaccination for up to 6 months post-vaccination.
Arm/Group | ACAM2000 Dose 1 | ACAM2000 Dose 2 | ACAM2000 Dose 3 | ACAM2000 Dose 4 | Dryvax® Vaccine
Serious Adverse Events (participants affected / at risk) | 1/51 | 1/102 | 0/102 | 0/50 | 0/52
Other Adverse Events (participants affected / at risk) | 48/51 | 93/102 | 98/102 | 49/50 | 51/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACAM2000 Dose 1 (N=51) | ACAM2000 Dose 2 (N=102) | ACAM2000 Dose 3 (N=102) | ACAM2000 Dose 4 (N=50) | Dryvax® Vaccine (N=52)
Pregnancy Not Otherwise Specified (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HIV test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ACAM2000 Dose 1 (N=51) | ACAM2000 Dose 2 (N=102) | ACAM2000 Dose 3 (N=102) | ACAM2000 Dose 4 (N=50) | Dryvax® Vaccine (N=52)
Lymph Node Pain (Blood and lymphatic system disorders) | 5 | 8 | 20 | 14 | 12
Lymphadenopathy (Blood and lymphatic system disorders) | 3 | 5 | 6 | 1 | 5
Diarrhea Not Otherwise Specified (Gastrointestinal disorders) | 8 | 17 | 11 | 12 | 9
Nausea (Gastrointestinal disorders) | 7 | 8 | 11 | 8 | 5
Constipation (Gastrointestinal disorders) | 4 | 5 | 9 | 3 | 3
Injection Site Pruritus (General disorders) | 29 | 59 | 77 | 38 | 43
Injection Site Erythema (General disorders) | 20 | 42 | 48 | 24 | 30
Fatigue (General disorders) | 15 | 28 | 41 | 18 | 18
Malaise (General disorders) | 17 | 20 | 29 | 18 | 15
Feeling Hot (General disorders) | 12 | 15 | 14 | 13 | 6
Rigors (General disorders) | 9 | 11 | 13 | 10 | 8
Injection Site Inflammation (General disorders) | 0 | 3 | 7 | 7 | 11
Injection Site Pain (General disorders) | 13 | 27 | 36 | 16 | 19
Myalgia (Musculoskeletal and connective tissue disorders) | 14 | 33 | 30 | 15 | 7
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 6 | 4 | 1 | 4
Headache Not Otherwise Specified (Nervous system disorders) | 24 | 39 | 46 | 25 | 21
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 7 | 2 | 2
Nasopharyngitis (Infections and infestations) | 1 | 1 | 11 | 7 | 3
Rash Not Otherwise Specified (Skin and subcutaneous tissue disorders) | 2 | 5 | 5 | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications